CLINICAL TRIAL: NCT06048406
Title: Effect of Health Education on Promoting Influenza Vaccination Health Literacy Among Primary School Students
Brief Title: Effect of Health Education on Promoting Influenza Vaccination Health Literacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Xu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SunYat-senU20230908
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Vaccination; Infection; Influenza
Keywords: health education; health literacy; schools; China
MeSH Terms: conditions — Infections; Influenza, Human; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will not know the intervention status of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a monthly health education intervention focused on influenza vaccination literacy for 5 months.
  Interventions: Combination Product: Health education
- Control (No Intervention): The control group will continue with their routine school health education for 5 months.

INTERVENTIONS:
Combination Product: Health education — The intervention group will receive a health education intervention focused on influenza vaccination literacy, while the control group will continue with their standard school health education without any additional intervention. An influenza vaccination health education including topics such as the importance of influenza vaccination, benefits of vaccination, and vaccination methods, will be developed and reviewed by an expert group. The package for the intervention group will include educational activities, distribution of promotional materials, vaccination services, and distribution of vaccination souvenirs.
  Arms: Intervention

SUMMARY:
The goal of this cluster randomized controlled trial is to evaluate the effect of health education interventions on influenza vaccination rates and health literacy in primary school students in the city of Dongguan in China.

Individuals aged 7 to 12 years who are in grades 4-5 in primary schools in Dongguan will be enrolled. 20 primary schools will be randomly selected, with half designated as intervention group schools and the remaining half as control group schools. The intervention group will receive a monthly health education intervention focused on influenza vaccination for 5 months, while the control group will continue with their routine school health education for 5 months.

Researchers will compare the differences in influenza vaccination rates and influenza vaccination health literacy levels between the intervention and control groups after 5 months to see if health education can promote influenza vaccination health literacy among primary school students.

DETAILED DESCRIPTION:
Introduction: Influenza is a major public health threat, and vaccination is the most effective prevention method. However, vaccination coverage remains suboptimal. Low health literacy regarding influenza vaccination may contribute to vaccine hesitancy. This study aims to evaluate the effect of health education interventions on influenza vaccination rates and health literacy.

Methods and analysis: This cluster randomized controlled trial will enroll 3036 students in grades 4-5 from 20 primary schools in Dongguan City, China. Schools will be randomized to an intervention group receiving influenza vaccination health education or a control group receiving routine health education. The primary outcome is influenza vaccination rate. Secondary outcomes include health literacy levels, influenza diagnosis rate, influenza-like illness incidence, and vaccine protection rate. Data will be collected through questionnaires, influenza surveillance, and self-reports at baseline and study conclusion.

Ethics and dissemination: Ethical approval has been sought from the Ethics Committee of the School of Public Health, Sun Yat-sen University. Findings from the study will be made accessible to both peer-reviewed journals and key stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Primary school students within the age range of 7-12 years.
* Students and their parents who voluntarily agree to participate in the study and provide signed informed consent.
* Permanent residents of Dongguan City who are expected to complete the project without transferring schools during the study period.

Exclusion Criteria:

* Individuals with contraindications to influenza vaccination, who have recently received an influenza vaccination, diagnosed with influenza or confirmed as influenza-like cases at the commencement of the study.
* Unwilling to participate in the project.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3036 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
influenza vaccination rate | Within 20 weeks from enrollment
  he influenza vaccination rate will be calculated as the number of vaccinated individuals divided by the total number of individuals, multiplied by 100%.

SECONDARY OUTCOMES:
influenza vaccination health literacy level | Within 20 weeks from enrollment
  Regarding the influenza vaccination health literacy level, each correct answer for the health literacy research questionnaire will be scored as one point, with incorrect answers receiving no points.
influenza incidence | Within 20 weeks from enrollment
  The influenza incidence will be calculated as the number of individuals diagnosed with influenza divided by the total number of individuals, multiplied by 100%
influenza vaccine protection rate | Within 20 weeks from enrollment
  The influenza vaccine protection rate will be calculated as the difference between the incidence rate in unvaccinated individuals and the incidence rate in vaccinated individuals, divided by the incidence rate in unvaccinated individuals, multiplied by 100%.
influenza-like illness incidence | Within 20 weeks from enrollment
  The ILI incidence will be calculated as the number of ILI cases divided by the total number of participants, multiplied by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Xu, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Dongguang Center for Disease Control and Prevention, Dongzhoucun, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Xie W, Huang X, Huang A, Lu T, Zhang R, Xiao J, He S, Wang J, Xu L. Impact of multifaceted health education on influenza vaccination health literacy in primary school students: a cluster randomized controlled trial. BMC Med. 2025 Jun 4;23(1):333. doi: 10.1186/s12916-025-04156-1. PMID 40468328
- [Derived] Xie W, Xiao J, Chen J, Huang H, Huang X, He S, Xu L. Impact of health education on promoting influenza vaccination health literacy in primary school students: a cluster randomised controlled trial protocol. BMJ Open. 2024 Apr 12;14(4):e080115. doi: 10.1136/bmjopen-2023-080115. PMID 38609315

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT06048406/Prot_SAP_000.pdf